CLINICAL TRIAL: NCT06421584
Title: Laparoscopic Cholecystectomy - A Randomized Controlled Trial Evaluating The Role Of Surgical Telementoring In Acquisition of Surgical Skills
Brief Title: Evaluating the Role of SURGical TElementoring in Acquisition of Surgical Skills of Laparoscopic Cholecystectomy. SURGTEACH Trial
Acronym: SURGTEACH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: Olympus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Nordlandssykehuset
Record Dates: First submitted 2024-04-11; First posted 2024-05-20 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-05

CONDITIONS: Surgical Education; Surgical Telementoring
Keywords: Competency based surgical education; Surgical telementoring; Laparoscopic cholecystectomy; Randomized controlled clinical trial

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial (RCT) was designed as a superiority trial to demonstrate the superiority of telementored resident skill learning in the operating room (OR) compared to standard training methods.
Who Masked: Participant, Outcomes Assessor
Masking Description: Mentors and telementors performing the GOALS-assessment of the video records are blinded to the temporal order of the performed procedures by the residents in both groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The residents randomized to the control arm will receive traditional intra operative guidance by the mentor holding the laparoscopic camera during the procedure.
- Interventional arm (Experimental): The residents randomized to the intervention arm will receive telementored guidance. This guidance is provided by telecommunication setup allowing the remotely located mentor to see the live footage of the laparoscopic procedure and to verbally communicate with the resident performing the surgical procedure.
  Interventions: Device: Surgical telementoring

INTERVENTIONS:
Device: Surgical telementoring — The intervention group receives intraoperative guidance by telementoring. The telementor is remotely located but able to see the real-time footage of the ongoing procedure and simultaneously verbally communicate with the operating resident wearing a headset during surgery. Additionally, feedback by telestration may be given to the operating resident if required. This involves graphic annotations on a still picture of the ongoing surgery which the telementor may design if required.
  Arms: Interventional arm

SUMMARY:
Surgical telementoring (ST) has the potential to become an integrated part of everyday surgical teaching practice. Its educational benefits require investigation.

This is a randomized controlled trial evaluating ST in a clinical setting. Laparoscopic cholecystectomy will be performed by eligible surgical residents randomized to the intervention group or the control group. The control group being guided by traditional onsite mentoring and the intervention group being telementored by a distantly located telementor during ongoing procedure. The primary outcome will be the video recorded GOALS-score (Global Operative Assessment of Laparoscopic Skills) and NOTSS-score (Non Technical Surgical Skills) assessment of each procedure while secondary outcomes will be satisfaction scores of the involved residents and mentors.

DETAILED DESCRIPTION:
Background:

Developing surgical skills among residents takes time and resources. Surgical practice is increasingly driven by efficacy and hospital economics. Operating room surgical education might conflict with these goals. The identified factors need optimizing surgical resident training. Surgical telementoring (ST) seems natural in surgery. Some ST-systems are cost-effective and safe. Despite recent technical breakthroughs and growing experience with telemedicine in the health sector, data on educational outcomes is still being determined.

Objective:

ST will be evaluated for efficiency and safety as a skill development tool for laparoscopic cholecystectomy. In this randomized controlled trial, surgical residents will be randomly assigned in a 1:1 ratio to the intervention group (real-time telementoring and postoperative coaching) or the control group (traditional intraoperative hands-on teaching). The research follows CONSORT, SPIRIT 2013 statements and the intention to treat principle (ITT).

The study is approved by the Norwegian ethical committee (REK HELSE NORD 32592) and the data protection officer (PVO) at Nordland Hospital trust Bodø (NLSH Bodø).

Two groups of residents will be allocated. The control group will follow the traditional hands-on surgical training method. In the intervention group, an expert surgeon will telementor the surgical residents. General surgery trainees in years 1-6 who have completed more than five laparoscopic abdominal surgeries are eligible. Stratification according to previous experience of the mentee will be made. All residents must agree with the mentor on surgical communication. This model uses LapcoNor principles for intraoperative communication and the GROW-model as an educational model. The GOALS score is the primary trial outcome. It consists of a five-item global rating scale for laparoscopic surgical skills. Each item may be scored from 1 to 5, where 1 is the lowest and five is the highest. The max score is 25. We hypothesize that the intervention group will enhance clinical skills by 3-5 points on the GOALS score compared to the control group. To attain 0.8 statistical power, a p-value of less than 0.05, and a 20% dropout rate, 12 residents per group are needed.

In addition to the GOALS-score assessment of video records, the NOTSS-score evaluating non-surgical technical skills will be assessed. The NOTSS score is based on 4 categories where each category consists of 3 elements. Each element may be graded from 1 to 4 , where 1 is the lowest and 4 is the highest. The highest achievable score is 48.

The higher the score, the better the outcome for both scoring systems.

Results:

Lapco TT courses were given to all telementors and onsite consulting surgeons before the trial start. In December 2023, the Medprescence (c) telementoring system was installed in three local hospitals. Residents, consultant surgeons, and telementors learned Medprescence setup and use. Surgical residents will be recruited once this research protocol is evaluated and accepted for publication to accommodate any necessary changes before the study begins. Starting recruitment in spring 2024 is feasible. This would allow data analysis by end of 2024 and publication in an international peer-reviewed journal by spring 2025.

Conclusions:

The SURGTEACH trial is the first randomized trial of telementoring for surgical education. The surgical education system and surgeon supply are limited globally and locally. Due to geographical and educational barriers, the Norwegian healthcare system requires support in educating enough surgeons. Therefore, surgical education must evolve, and surgical telementoring may help solve these challenges. This research may give high quality evidence to improve surgical education, especially in rural hospitals.

ELIGIBILITY:
Inclusion criteria for residents in control- and intervention group:

* General surgery residents in years 1 to 6 of their specialty education having performed more than five laparoscopic procedures.
* Stratification according to experience will be made for the subject in the control arm and in the intervention arm.
* Having passed the prerequisite mandatory national course of general laparoscopic principles.
* All residents had to undergo agreement with the mentor about communication model during surgery. This model is derived from LapcoNor principals (11). Residents in the intervention group underwent an additional introduction to the principals of communication through telementoring at the OR. They were introduced to the telementoring equipment.

Inclusion criteria for on-site mentors (control group) and telementors (intervention group): • - Consultant surgeon with more than 3 years of experience with independently performing laparoscopic cholecystectomies.

* Having acquaintance with assessment of videos for GOALS-score (12)
* Both telementors and on-site mentors had to show certificate of having done the national LapCo-Nor "train the trainer" course and followed standardized norms of communication with the mentee during surgical mentoring thus diminishing bias of communicative difference.

Inclusion criteria for included patients:

* Gallstone disease without clinical history of cholecystitis
* BMI < 38
* No previous history of upper abdominal laparotomy
* No previous history of percutaneous gallbladder drainage
* Patient provided informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
GOALS-score (Global Operative Assessment of Laparoscopic Skills) | Each resident in both the intervention group and the control group will be scheduled to perform 5 consecutive laparoscopic cholecystectomies within 3-5 days.
  GOALS-score is a validated scoring system for laparoscopic surgical skills. Each performed procedure in the control group and the intervention group will be divided into 5 key-steps and each step will be scored by the 5 involved mentors and telementors. The video records of the procedures will be edited by the main author into 5 key-steps. Each recorded procedure will not exceed 1hours duration. All five procedures by each resident will be edited and presented to 5 mentors/telementors for GOALS-score assessment. Total GOALS-score will be calculated by adding the scores of each key-step.
  Every resident in each of the 2 groups will perform 5 consecutive procedures within 3-5 consecutive days. The GOALS-assessment will be required with 1 week after presenting the procedures to the 5 mentors/telementors
NOTSS-score (Non-technical surgical skills) | Each resident in both the intervention group and the control group will be scheduled to perform 5 consecutive laparoscopic cholecystectomies within 3-5 days.
  Assessing non-surgical technical skills by assessment of 4 categories (Situation awareness, Decision making, Communication and teamwork and Leadership. Each category consists of 3 elements. Each category is rated from 1-4 and each of the 3 elements within each category is rated from 1-4. Each recorded and edited video record of the 5 consecutive laparoscopic procedures by the residents in both groups will be presented to mentors/telementors (5 members) for NOTSS-score assessment. The NOTSS-assessment will be required with 1 week after presenting the procedures to the 5 mentors/telementors.

SECONDARY OUTCOMES:
Satisfaction score of residents in the control group and the intervention group. | 5 subsequent procedures will be performed by each resident within a periode of 3-5 days. Satisfaction score form will be asked for within 1 hour after each procedure.
  Each resident (both groups) will be given a predetermined form for self-reported satisfaction score. Resident satisfaction survey was based on a 5-point Likert scale. 7 statements are to be assessed with answers ranging from 1= strong disagreement with the statement and 5=strong agreement with the statement. 5 is the best outcome for each statement and 35 is the best overall result for the survey.
Satisfaction score of mentors (control group) and telementors (intervention group) | Each mentor and telementor will be given a satisfaction score form to fill out within 1 hour after each procedure.
  Each mentor and telementor (both groups)will be given a predetermined form for self-reported satisfaction score. The mentor/telementor satisfaction survey was based on a 5-point Likert scale. 7 statements are to be assessed with answers ranging from 1= strong disagreement with the statement and 5=strong agreement with the statement. 5 is the best outcome for each statement and 35 is the best overall result for the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Petter Øien, PhD, Study Director — Head of research department
Locations (1):
- NordlandssykehusetHF, Bodø, Nordland, Norway

IPD SHARING:
Plan to Share IPD: Yes
Video records of the procedures will be stripped for patient-ID and stored anonymously on a secured website. Each video will be given an URL-address. The study secretary will have the key enabling recognition of each video to the specific patient and performing surgeon. The anonymous video records will be made available for each of the 5 mentors/telementors after being edited and labelled with key-steps of the procedure. Blinded GOALS- and NOTSS-assessment by the mentors/telementors will be performed. The assessment results will be collected by the study secretary on a questback scheme handed out in advance to the evaluators. The study secretary possesses the key enabling recognition of the video records according to patient-ID and performing residents. An Excel file with the results will be constructed by the study secretary and the data analysis will be commenced. The video records and the Excel file, constituting the raw data, will be available as IPD for sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available as it is collected. Videorecords of the procedures by the residents are planned to be finished by end of November 2024. The video records will be stored continuously and the website will be availabe at the starting point. The GOALS-scores and NOTSS-scores will be collected continuously as the video records are edited and presented to the mentors (control arm) and the telementors (intervention arm)
Access Criteria: All raw data will be shared on request.

REFERENCES:
- [Background] Holmer H, Lantz A, Kunjumen T, Finlayson S, Hoyler M, Siyam A, Montenegro H, Kelley ET, Campbell J, Cherian MN, Hagander L. Global distribution of surgeons, anaesthesiologists, and obstetricians. Lancet Glob Health. 2015 Apr 27;3 Suppl 2:S9-11. doi: 10.1016/S2214-109X(14)70349-3. No abstract available. PMID 25926323
- [Background] Vickers AJ, Bianco FJ, Gonen M, Cronin AM, Eastham JA, Schrag D, Klein EA, Reuther AM, Kattan MW, Pontes JE, Scardino PT. Effects of pathologic stage on the learning curve for radical prostatectomy: evidence that recurrence in organ-confined cancer is largely related to inadequate surgical technique. Eur Urol. 2008 May;53(5):960-6. doi: 10.1016/j.eururo.2008.01.005. Epub 2008 Jan 14. PMID 18207316
- [Background] Zorn KC, Gautam G, Shalhav AL, Clayman RV, Ahlering TE, Albala DM, Lee DI, Sundaram CP, Matin SF, Castle EP, Winfield HN, Gettman MT, Lee BR, Thomas R, Patel VR, Leveillee RJ, Wong C, Badlani GH, Rha KH, Eggener SE, Wiklund P, Mottrie A, Atug F, Kural AR, Joseph JV; Members of the Society of Urologic Robotic Surgeons. Training, credentialing, proctoring and medicolegal risks of robotic urological surgery: recommendations of the society of urologic robotic surgeons. J Urol. 2009 Sep;182(3):1126-32. doi: 10.1016/j.juro.2009.05.042. Epub 2009 Jul 21. PMID 19625032
- [Background] Strasberg SM, Hertl M, Soper NJ. An analysis of the problem of biliary injury during laparoscopic cholecystectomy. J Am Coll Surg. 1995 Jan;180(1):101-25. No abstract available. PMID 8000648
- [Background] Yun Kyung Jung et al: What is the safe training to educate the laparoscopic cholecystectomy for surgical residents in early learning curve ? J. Minim Invasive Surg 2016; 19(2): 70-74
- [Background] Doarn CR. Telemedicine in tomorrow's operating room: a natural fit. Semin Laparosc Surg. 2003 Sep;10(3):121-6. doi: 10.1177/107155170301000305. PMID 14551654
- [Background] Ohinmaa A, Vuolio S, Haukipuro K, Winblad I. A cost-minimization analysis of orthopaedic consultations using videoconferencing in comparison with conventional consulting. J Telemed Telecare. 2002;8(5):283-9. doi: 10.1177/1357633X0200800507. PMID 12396857
- [Background] Schulam PG, Docimo SG, Saleh W, Breitenbach C, Moore RG, Kavoussi L. Telesurgical mentoring. Initial clinical experience. Surg Endosc. 1997 Oct;11(10):1001-5. doi: 10.1007/s004649900511. PMID 9381336
- [Background] Augestad KM, Bellika JG, Budrionis A, Chomutare T, Lindsetmo RO, Patel H, Delaney C; Mobile Medical Mentor (M3) Project. Surgical telementoring in knowledge translation--clinical outcomes and educational benefits: a comprehensive review. Surg Innov. 2013 Jun;20(3):273-81. doi: 10.1177/1553350612465793. Epub 2012 Oct 30. PMID 23117447
- [Background] Wood D. No surgeon should operate alone: how telementoring could change operations. Telemed J E Health. 2011 Apr;17(3):150-2. doi: 10.1089/tmj.2011.9986. No abstract available. PMID 21500973
- [Background] Hanna GB, Mackenzie H, Miskovic D, Ni M, Wyles S, Aylin P, Parvaiz A, Cecil T, Gudgeon A, Griffith J, Robinson JM, Selvasekar C, Rockall T, Acheson A, Maxwell-Armstrong C, Jenkins JT, Horgan A, Cunningham C, Lindsey I, Arulampalam T, Motson RW, Francis NK, Kennedy RH, Coleman MG; on behalfofLapco program. Laparoscopic Colorectal Surgery Outcomes Improved After National Training Program (LAPCO) for Specialists in England. Ann Surg. 2022 Jun 1;275(6):1149-1155. doi: 10.1097/SLA.0000000000004584. Epub 2020 Oct 19. PMID 33086313
- [Background] Vassiliou MC, Feldman LS, Andrew CG, Bergman S, Leffondre K, Stanbridge D, Fried GM. A global assessment tool for evaluation of intraoperative laparoscopic skills. Am J Surg. 2005 Jul;190(1):107-13. doi: 10.1016/j.amjsurg.2005.04.004. PMID 15972181
- [Background] Mackenzie H, Cuming T, Miskovic D, Wyles SM, Langsford L, Anderson J, Thomas-Gibson S, Valori R, Hanna GB, Coleman MG, Francis N. Design, delivery, and validation of a trainer curriculum for the national laparoscopic colorectal training program in England. Ann Surg. 2015 Jan;261(1):149-56. doi: 10.1097/SLA.0000000000000437. PMID 24374538
- [Background] Manatakis DK, Antonopoulou MI, Tasis N, Agalianos C, Tsouknidas I, Korkolis DP, Dervenis C. Critical View of Safety in Laparoscopic Cholecystectomy: A Systematic Review of Current Evidence and Future Perspectives. World J Surg. 2023 Mar;47(3):640-648. doi: 10.1007/s00268-022-06842-0. Epub 2022 Dec 6. PMID 36474120
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542